CLINICAL TRIAL: NCT03625622
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate Efficacy and Safety of 26-Week Treatment of AR1001 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety of 26-Week Treatment of AR1001 in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AriBio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR1001-ADP2-US01
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Mild to Moderate Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: After the first 26 weeks, subjects can participate in an optional extension study to receive either 10 mg or 30 mg AR1001 for another 26 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind for study site and participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, orally administered once daily for 26 weeks.
  Interventions: Drug: Placebo
- AR1001 - 10 mg (Active Comparator): Active, AR1001 - 10 mg, orally administered once daily for 26 weeks.
  Interventions: Drug: AR1001
- AR1001 - 30 mg (Active Comparator): Active, AR1001 - 30 mg, orally administered once daily for 26 weeks.
  Interventions: Drug: AR1001

INTERVENTIONS:
Drug: AR1001 — AR1001 Active Oral Tablet
  Arms: AR1001 - 10 mg; AR1001 - 30 mg
Drug: Placebo — Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
A double-blinded, randomized, placebo-controlled study will be performed to evaluate the efficacy and safety of treating AR1001 in patients with mild to moderate Alzheimer's disease for 26 weeks.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is the most prevalent neurodegenerative disorder in The United States affecting approximately 5.4 million Americans. AD is characterized by progressive loss in memory and as well as a decline in the ability to learn that is associated with neuronal death. Well known hallmarks of AD are neuritic plaques and neurofibrillary tangles and extensive inflammation. Currently, no treatment has been developed to fully cure or prevent the progression of dementia that is associated with AD.

AR1001 is a polypharmacological drug candidate being developed as a treatment for AD and shows great potential with favorable attributes for a central nervous system (CNS) drug (i.e., high specificity and potency, as well as good pharmacokinetic, bioavailability, CNS penetration, and ensured safety).

The clinical study of AR1001 aims to evaluate the efficacy and safety of AR1001 as a potential treatment for AD. Based on the preclinical results, AR1001 could be an effective treatment option with a mechanism of action that has not been explored for AD indication.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects aged 55-80 years at the time of signing the Informed Consent Form.
2. Subjects (or subject's legally acceptable representative) and caregiver(s) who can sign an Informed Consent to participate in the study. Same caregiver(s) must assist the subject throughout the entire duration of the study.
3. Subjects who have a diagnosis of probable Alzheimer's disease according to the NIA-AA (National Institute of Aging and Alzheimer's Associations, 2011) criteria with mild to moderate dementia (stage 4 - 5) at screening.
4. Subjects who have mild-to-moderate cognitive impairment with MMSE Score of 16-26 at screening.
5. Subjects who have an MRI (either 1.5T or 3T) or CT scan performed after onset of symptoms and prior to randomization with findings consistent with the diagnosis of dementia due to Alzheimer's disease and without any other clinically significant comorbid pathologies.
6. Subjects who have one (or more) identified adult study partner(s) who, in the opinion of the investigator, has sufficient contact with and knowledge about the subject as to be able to report knowledgeably about the subject's safety, compliance and adherence, cognition, function, and behavior.

Exclusion Criteria

1. Subjects who are female who are pregnant, nursing, or of childbearing potential and not practicing effective contraception.
2. Subjects who have signs of delirium.
3. Subjects who have had a cortical stroke within the preceding 2 years.
4. Subjects who have any diagnosis of dementia other than that related to Alzheimer's Disease, including concomitant vascular dementia.
5. Subjects who have a PET scan performed after onset of symptoms with negative amyloid results.
6. Subjects with a history of myocardial infarction, unstable angina, New York Heart Association (NYHA) class III or IV heart failure or stroke within the last 12 months.
7. Subjects with uncontrolled hypertension (systolic blood pressure >160mm Hg or diastolic blood pressure > 95mm Hg) or hypotension (systolic blood pressure <90mm Hg or diastolic blood pressure <50mm Hg).
8. Subjects who have clinically significant renal impairment (creatinine > 1.5x ULN) or hepatic impairment (AST or ALT > 2.5x ULN or total bilirubin > 1.5x ULN).
9. Subjects who have history of cancer or malignant tumor within 5 years prior to screening with the exception of:

   1. Basal or squamous cell carcinoma of the skin or cervical dysplasia which has been adequately treated.
   2. In situ Grade 1 cervical cancer, fully treated at least 2 years prior to screening and without recurrence.
   3. Prostate cancer, confined to the prostate gland, which has been adequately treated (surgery and/or radiation) with normal or low and stable PSA levels for 2 years prior to screening.
10. Subjects who have history of untreated thyroid disorder or a seizure disorder.
11. Subjects who are being treated, or likely to require treatment during the study, with any medications prohibited by the study protocol.
12. Subjects who have participated in any investigational drug or device trial within the previous 30 days or five half-lives of the investigational drug at screening, whichever one is longer.
13. Subjects who have any other clinically significant abnormal result in laboratory tests such as abnormally low B12 or high TSH levels, as determined by the Investigator.
14. Subjects with any current psychiatric diagnosis other than AD if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessments, or affect the subject's ability to complete the study.
15. Subjects whose treatment with FDA-approved AD medication (donepezil, galantamine, memantine, rivastigmine or their combinations) has not been stable for at least 3 months prior to screening. Treatment and dosing should remain stable, with no changes throughout the trial.
16. Subjects who are currently receiving (or unable to stop use for at least 21 days [3 weeks] prior to receiving the first dose of the AR1001 and throughout the study) prescription or non-prescription medications or other products known to be moderate or potent inhibitors/inducers of CYP3A4.
17. Subjects who have had any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the AR1001 and throughout the study.
18. Subjects, in the opinion of the Investigator, who are unsuitable to participate in the study.

Extension Phase Continuation Criterion

1. Subjects enrolled in AR1001-ADP2-US01 and completed 26 weeks of assigned dosing.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
ADAS-Cog 13 | 26 weeks
  Change of ADAS-Cog (Alzheimer's Disease Assessment Scale-cognitive subscale) from baseline at Week 26
ADCS-CGIC | 26 weeks
  Change of ADCS-CGIC (Alzheimer's disease Cooperative Study-Clinical Global Impression of Change)

SECONDARY OUTCOMES:
MMSE-2 | 26 weeks
  Change of MMSE (Mini-mental status examination) from baseline at Week 26
NPI | 26 weeks
  Changes of NPI (Neuropsychiatric Inventory) from baseline at Week 26
GDS | 26 weeks
  Changes of GDS (Geriatric Depression Scale) from baseline at Week 26
C-SSRS | 26 weeks
  Changes of C-SSRS (Columbia Suicide Severity Rating Scale) from baseline at Week 26
QOL-AD | 26 weeks
  Changes of QOL-AD (Quality of Life in Alzheimer's Disease) from baseline at Week 26
Treatment related adverse events | 26 weeks
  Number of subjects with treatment related adverse events as assessed by analysis of adverse events including symptoms and abnormal findings on physical examination, vital signs, ECG, and standard laboratory examination results

CONTACTS AND LOCATIONS:
Overall Officials: James Rock, Study Director — SVP of global development
Locations (21):
- United States (21):
  - Advanced Clinical Research, Inc., Banning, California
  - Northern California Research, Sacramento, California
  - Syrentis Clinical Research, Santa Ana, California
  - Meridien Research, Lakeland, Florida
  - Meridien - Maitland, Maitland, Florida
  - The Neurology Research Group, Miami, Florida
  - Accelerated Enrollment Solutions (AES), Orlando, Florida
  - IMIC, Inc, Palmetto Bay, Florida
  - Meridien Research - Spring Hill, Spring Hill, Florida
  - Meridien Research - St Petersburg, St. Petersburg, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - NeuroStudies, LLC, Decatur, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Wake Research - CRCNV, Las Vegas, Nevada
  - Rapid Medical Research, Beachwood, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Palmetto Clinical Research, Summerville, South Carolina
  - Advanced Clinical Research - Cedar Park, Cedar Park, Texas
  - FMC Science, Lampasas, Texas
  - Advanced Clinical Research, Inc., West Jordan, Utah
  - Kingfisher Cooperative, LLC, Spokane, Washington

REFERENCES:
- [Derived] Greeley D, Nash M, Herskowitz B, Kim F, Rock J, Prins N, Kim S, Xi T, Busam JA, Tete B, Choung JJ, Sha SJ. A phase 2 randomized, placebo-controlled study on the efficacy and safety of AR1001, a phosphodiesterase-5 inhibitor, in patients with mild-to-moderate Alzheimer's disease. J Prev Alzheimers Dis. 2025 Nov;12(9):100337. doi: 10.1016/j.tjpad.2025.100337. Epub 2025 Sep 5. PMID 40912996